CLINICAL TRIAL: NCT03785990
Title: Untersuchung Intraoperativ Entnommener Subkutaner Fettgewebeproben Früh- Und Reifgeborener Auf Die Fettsäure-Zusammensetzung Der Triglyceride Und Der Phospholipide Mit Speziellem Fokus Auf Die Mehrfach ungesättigten Fettsäuren Docosahexaensäure Und Arachidonsäure Wissenschaftliche Untersuchung Bei Minderjährigen
Brief Title: Fatty Acid Composition of Subcutaneous Adipose Tissue in Infants: A Prospective and Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-Adipose tissue
Record Dates: First submitted 2018-05-09; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-05

CONDITIONS: Prematurity; Subcutaneous Adipose Tissue
Keywords: preterm; fatty acid; docosahexaenoic acid; arachidonic acid; infant; adipose tissue; subcutaneous adipose tissue
MeSH Terms: conditions — Premature Birth | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- preterms with enterostomy: GA 23±0/7 - 31±6/7 with clinically indicated operations because of NEC (necrotising enterocolitis) or FIP (focal intestinal perforation). Operation after birth (within 14 days) and at term (enterostomy closure) Analysis of the blood, subcutaneous adipose tissue und total adipose tissue (PEAPOD)
  Interventions: Other: adipose tissue; Other: blood; Diagnostic Test: PEAPOD
- preterms without enterostomy: GA 23±0/7 bis 31±6/7 with a clinically indicated operation (e.g. herniotomy) at term, without any abdominal problems.
  Analysis of the blood, subcutaneous adipose tissue und total adipose tissue (PEAPOD)
  Interventions: Other: adipose tissue; Other: blood; Diagnostic Test: PEAPOD
- term infants: GA ≥34±0/7 with a clinically indicated operation directly after birth (within 14 days) (e.g. gastroschisis).
  Analysis of the blood, subcutaneous adipose tissue und total adipose tissue (PEAPOD)
  Interventions: Other: adipose tissue; Other: blood; Diagnostic Test: PEAPOD

INTERVENTIONS:
Other: adipose tissue — taking a sample of the adipose tissue during operation
Other: blood — taking a blood sample when a peripheral venous catheter is inserted before operation
Diagnostic Test: PEAPOD — Measurement of the total adipose tissue of the infant with PEAPOD (Air Displacement-Plethysmography, Infant Body Composition System, Cosmed, Rome, Italy)

SUMMARY:
The fatty acid composition in blood and subcutaneous adipose tissue of infants that have an clinical indicated operation is studied.

DETAILED DESCRIPTION:
Collection of:

* subcutaneous adipose tissue of term infants and preterms after birth and at term during a clinically indicated operation.
* blood before the operation.

Measurement of the fatty acid composition (especially arachidonic acid and docosahexaenoic acid) in subcutaneous adipose tissue and blood.

Aim is to compare the composition of the fatty acids in blood and adipose tissue of preterms at term and term infants. To calculate the fatty acid value in each infant the proportion of adipose tissue is determined with PEAPOD before discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* meeting criteria of the 3 cohorts

Exclusion Criteria:

* metabolic diseases of the infant
* genetic diseases
* missing agreement for the study

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: term and preterm neonates
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Fatty acid composition of the subcutaneous adipose tissue and plasma | at the time of the operation
  Fatty acid composition of the subcutaneous adipose tissue and plasma of preterms at term compared to the composition of infants after birth (within 14 days).

SECONDARY OUTCOMES:
Fatty acid composition of the subcutaneous adipose tissue and plasma of preterms with abdominal problems | time of the first operation until discharge home (at a postnatal age of up to 4-5 months at the most in very preterm infants)
  Change of fatty acid composition of the subcutaneous tissue and plasma from first to second operation in preterms with abdominal operations, enterostomy
Fatty acid composition of the subcutaneous adipose tissue and plasma of preterms with abdominal problems and preterms without abdominal problems at term | time of the first operation until discharge home (at a postnatal age of up to 4-5 months at the most in very preterm infants)
  Fatty acid composition of the subcutaneous adipose tissue and plasma of preterms at term compared to the composition of preterms at term with enterostomy.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bockmann KA, von Stumpff A, Bernhard W, Shunova A, Minarski M, Frische B, Warmann S, Schleicher E, Poets CF, Franz AR. Fatty acid composition of adipose tissue at term indicates deficiency of arachidonic and docosahexaenoic acid and excessive linoleic acid supply in preterm infants. Eur J Nutr. 2021 Mar;60(2):861-872. doi: 10.1007/s00394-020-02293-2. Epub 2020 May 31. PMID 32476053